CLINICAL TRIAL: NCT00829842
Title: Evaluation of Oral Hygiene With 0.12% Chlorhexidine Antiseptic Solution on the Incidence of Nosocomial Pneumonia and Ventilator-Associated Pneumonia in Children Submitted to Heart Surgery
Brief Title: Oral Hygiene With Chlorhexidine and Incidence of Ventilator-Associated Pneumonia in Children Submitted to Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HCRP 8904/2005
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Ventilator Associated Pneumonia; Nosocomial Pneumonia; Heart Surgery
Keywords: chlorexidine; ventilator-associated pneumonia; nosocomial pneumonia; heart surgery; oral hygiene
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia | interventions — Oral Hygiene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Other: placebo
- 2 (Experimental)
  Interventions: Other: oral hygiene

INTERVENTIONS:
Other: oral hygiene — oral hygiene with 0.12% chlorexidine
  Arms: 2
Other: placebo — oral hygiene placebo
  Arms: 1

SUMMARY:
Hospital infections play an important role in the increase of patients' morbimortality and hospitalization costs, especially in the case of individuals admitted to intensive care units (ICU) during postoperative heart surgery. Analysis of the epidemiological profile of the hospital infections in the pediatric-ICU (P-ICU) of Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, University of São Paulo (HCFMRP-USP) demonstrated a 31.1% incidence of pneumonia (PNM) and a rate of ventilator-associated pneumonia (VAP) of 23.81 per 1000 ventilators-day between March 2004 and February 2005 in the group submitted to cardiac surgery. Knowledge of the pathophysiology and risk factors associated with this infection allows for measures aiming at reducing its incidence. The objective of the present study is to evaluate the effect of oral hygiene with a 0.12% chlorhexidine solution on the incidence of PNM and PAV in children submitted to cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 0 to 18 years submitted to heart surgery
* parent approval

Exclusion Criteria:

* previous oral intubation
* previous or present pneumonia
* parent refusal
* death during surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2006-02; Study Completion 2006-02 (Actual)

REFERENCES:
- [Derived] Jacomo AD, Carmona F, Matsuno AK, Manso PH, Carlotti AP. Effect of oral hygiene with 0.12% chlorhexidine gluconate on the incidence of nosocomial pneumonia in children undergoing cardiac surgery. Infect Control Hosp Epidemiol. 2011 Jun;32(6):591-6. doi: 10.1086/660018. PMID 21558772